CLINICAL TRIAL: NCT01834313
Title: Identifying Patients' and Healht Insurers' Preferences Regarding Patient-centred Care by Determining Their Willingness-to-pay for Patient-centred Care
Brief Title: Willingness to Pay for Patient-centred Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A.G. Huppelschoten (Other)
Responsible Party: Sponsor-Investigator, A.G. Huppelschoten, MD, Principal Investigator, University Medical Center Nijmegen
Organization: University Medical Center Nijmegen (Other)
Other Study IDs: DCE
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Willingness-to-pay; Patient-centredness
Keywords: Willingness-to-pay; Patient-centredness; Health insurers; Fertility care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the monetary value of patient-centrednes in health care by determining a willingness-to-pay for more patient-centredness care for both patients and health insurers

DETAILED DESCRIPTION:
We perform our study in the area of fertility care, as it is known that infertile patients suffer from a high physical and physiological burden during treatment and could especially benefit from patient-centred care. Moreover, previous studies have clearly identified the concept of patient-centred fertility care and have shown that improvement is needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing MAR-treatment (ovulation induction, intra-uterine inseminations, in vitro fertilization, or intra-cytoplasmic sperm injection)
* All healthcare purchasers working at one of the 5 large Dutch health insurer companies.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who are under treatment for their fertility problem and underwent at least one treatment in one of 10 Dutch clinics.
  All healthcare purchasers from the 5 large Dutch health insurer companies
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-08 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Willingness-to-pay for patient-centred care | 6 months
  A willingness-to-pay for patient-centred care for both patients and health insurers

CONTACTS AND LOCATIONS:
Overall Officials: J AM Kremer, MD, PhD, Study Chair — Radboud University Medical Centre, Nijmegen; W L Nelen, MD, PhD, Study Director — Radboud University Medical Centre, Nijmegen; E MM Adang, PhD, Study Director — Radboud University Medical Centre, Nijmegen; A G Huppelschoten, MD, Principal Investigator — Radboud University Medical Centre, Nijmegen
Locations (1):
- Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Huppelschoten AG, Verkerk EW, Appleby J, Groenewoud H, Adang EM, Nelen WL, Kremer JA. The monetary value of patient-centred care: results from a discrete choice experiment in Dutch fertility care. Hum Reprod. 2014 Aug;29(8):1712-20. doi: 10.1093/humrep/deu122. Epub 2014 Jun 4. PMID 24903199